CLINICAL TRIAL: NCT06550700
Title: The Outcomes of Simultaneous Resection for Colorectal Cancer Liver Metastases by Laparoscopic Hybrid Surgery Versus Totally Open Surgery: a Prospective Cohort Study
Brief Title: The Outcomes of Laparoscopic Hybrid Surgery Versus Totally Open Surgery
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Department of Colorectal Surgery, Changhai Hospital
Other Study IDs: CHLM
Record Dates: First submitted 2024-06-19; First posted 2024-08-13 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Resectable Simultaneous Colorectal Cancer Liver Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic hybrid surgery (LHS) cohort: Routine colorectal surgery is performed first, followed by liver surgery. The LHS cohort first performed the laparoscopic exploration of the entire abdominal-pelvic cavity to determine the resectability of the primary and metastatic lesions. After the blood vessel detachment and bowel detachment, the distal bowel of the tumor was severed and the pneumoperitoneum was closed. The liver metastases were then removed in both cohorts by open resection through the right subcostal incision.
  Interventions: Procedure: laparoscopic hybrid surgery (LHS)
- totally open surgery (TOS) cohort: Routine colorectal surgery is performed first, followed by liver surgery. The blood vessel detachment, bowel detachment, the distal bowel of the tumor in the TOS cohort were accomplished by open surgery through the mid-abdominal incision approach. The liver metastases were then removed in both cohorts by open resection through the right subcostal incision.

INTERVENTIONS:
Procedure: laparoscopic hybrid surgery (LHS) — First performed the laparoscopic exploration of the entire abdominal-pelvic cavity to determine the resectability of the primary and metastatic lesions. After the blood vessel detachment and bowel detachment, the distal bowel of the tumor was severed and the pneumoperitoneum was closed. The liver metastases were then removed in both cohorts by open resection through the right subcostal incision.
  Groups: laparoscopic hybrid surgery (LHS) cohort

SUMMARY:
Simultaneous colorectal cancer liver metastasis (SCRLM) is one of the risk factors for poor prognosis in colorectal cancer. Surgical resection of primary and metastatic lesions is the first choice of treatment for patients with resectable SCRLM. Simultaneous resection of colorectal cancer liver metastases by totally open surgery (TOS) has been widely used. However, we propose that laparoscopic hybrid surgery (LHS) may have better short and long-term outcomes. This study aimed to compare the safety, short-term, and long-term efficacy of LHS versus TOS for patients with resectable SCRLMs.

ELIGIBILITY:
Inclusion Criteria:

* Liver metastasis was detected while the colorectal cancer was diagnosed.
* Both the primary lesions and liver metastases were confirmed by postoperative pathological examination.
* Clinical data is complete.

Exclusion Criteria:

* Patients with unresectable extrahepatic metastases.
* Patients with other malignant tumor diseases that have not been cured.
* Clinical and pathological data were missed or incomplete follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study collected clinical data from patients who underwent simultaneous resection of colorectal cancer liver metastases at the Department of Colorectal Surgery in Changhai Hospital from January 2010 to June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
short-term outcome: Operative time | Within one week of the patient undergoing surgery
  Time taken for surgery
short-term outcome: Blood loss | Within one week of the patient undergoing surgery
  Patient haemorrhage during surgery
short-term outcome: Time of liquid diet | Within one week of the patient undergoing surgery
  Time for patients to eat fluids for the first time after surgery
short-term outcome: Postoperative hospital stay | Within one week of the patient undergoing surgery
  Length of stay of patients after surgery
short-term outcome: Surgical complications | Within one week of the patient undergoing surgery
  Complications that occur in patients after surgery

SECONDARY OUTCOMES:
overall survival (OS) | 3years
  the time after surgical treatment until death for any reason
disease-free survival (DFS) | 3years
  the time after surgical treatment until the first observation of tumor recurrence or death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No